CLINICAL TRIAL: NCT01467570
Title: Efficacy and Safety of a New Oral Rehydration Solution (Hipp ORS 200 Apple) in Children With Acute Gastroenteritis: Randomized, Double-Blind Controlled Trial
Brief Title: Efficacy and Safety of a New Oral Rehydration Solution (Hipp ORS 200 Apple) in Children With Acute Gastroenteritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB/191/2008
Record Dates: First submitted 2011-10-27; First posted 2011-11-08 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2013-11

CONDITIONS: Diarrhea
Keywords: diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hipp ORS Apple 200 (Experimental): oral rehydration solution Hipp ORS 200 Apple
  Interventions: Dietary Supplement: oral rehydration solution Hipp ORS Apple 200
- ESPGHAN ORS (Active Comparator): ESPGHAN oral rehydration solution
  Interventions: Dietary Supplement: ESPGHAN ORS

INTERVENTIONS:
Dietary Supplement: oral rehydration solution Hipp ORS Apple 200 — Volume of the solution calculated by weight:
  * fast oral rehydration in 3-4 hours by mouth
  * ORS given for ongoing losses until diarrhea stops (maintenance phase)
  Arms: Hipp ORS Apple 200
Dietary Supplement: ESPGHAN ORS — Volume of the solution calculated by weight:
  * fast oral rehydration in 3-4 hours by mouth
  * ORS given for ongoing losses until diarrhea stops (maintenance phase)
  Arms: ESPGHAN ORS

SUMMARY:
It is generally recommended that oral rehydration should be used as first-line therapy to treat or prevent dehydration in children with acute gastroenteritis (AGE). Refusal to drink regular Oral Rehydration Solution (ORS) interfere with compliance with the recommended treatment.

The objective of this study is to compare the tolerance, acceptance, efficacy and safety of a new ORS (Hipp ORS 200 Apple) of improved palatability with regular ORS recommended by ESPGHAN in children with acute gastroenteritis (AGE).

DETAILED DESCRIPTION:
It is generally recommended that oral rehydration should be used as first-line therapy to treat or prevent dehydration in children with acute gastroenteritis (AGE). Despite the proven efficacy of oral rehydration therapy it remains underused. The main reason for this is that an ORS neither reduces the frequency of bowel movements and fluid loss nor shortens the duration of illness, which decreases its acceptance. Moreover, unpalatability of regular ORS decrease its acceptance, especially in children with lower degrees of dehydration. Refusal to drink regular ORS interfere with compliance with the recommended treatment. Parents, but also health care professionals, demand safe, effective, inexpensive, but also well tolerated and accepted ORS for management of AGE.

Recently, a new ORS (Hipp ORS 200 Apple) with improved taste has been developed, and is now frequently employed for the management of AGE. The proposed study will be the first double-blind randomized trial of this ORS. It will evaluate clinically meaningful benefits to be derived by children and caregivers from its use. If positive, this new ORS may become a routine recommendation for children with AGE.

The objective of this study is to compare the tolerance, acceptance, efficacy and safety of a new ORS (Hipp ORS 200 Apple) with regular ORS recommended by ESPGHAN in children with AGE.

ELIGIBILITY:
Inclusion Criteria:

* children age 4 to 48 months
* diarrhoea defined as the passage of three or more loose or watery stools per day for >1 but <5 days
* mild (3%) or moderate dehydration (3-9%) according to the World Health Organization criteria (Table 1)
* informed consent signed by at least one parent / caregiver

Exclusion Criteria:

* diarrhea for <1 or >5 days
* severe dehydration (>9%)
* recent history of diarrhea indicated either by parent/guardian or hospital case notes
* underlying chronic gastrointestinal disease (i.e., celiac disease, cow's milk protein intolerance)
* breastfeeding >50%
* under nutrition (weight/height ratio below the fifth percentile)
* systemic infections
* immune defects or immunosuppressive treatment

Ages: 4 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hania Szajewska, Professor, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Peadiatrics, The Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Background] Guarino A, Albano F, Ashkenazi S, Gendrel D, Hoekstra JH, Shamir R, Szajewska H; ESPGHAN/ESPID Evidence-Based Guidelines for the Management of Acute Gastroenteritis in Children in Europe Expert Working Group. European Society for Paediatric Gastroenterology, Hepatology, and Nutrition/European Society for Paediatric Infectious Diseases evidence-based guidelines for the management of acute gastroenteritis in children in Europe: executive summary. J Pediatr Gastroenterol Nutr. 2008 May;46(5):619-21. doi: 10.1097/MPG.0b013e31816e219e. No abstract available. PMID 18493225
- [Background] Recommendations for composition of oral rehydration solutions for the children of Europe. Report of an ESPGAN Working Group. J Pediatr Gastroenterol Nutr. 1992 Jan;14(1):113-5. No abstract available. PMID 1573500
- [Background] Szajewska H, Hoekstra JH, Sandhu B; ESPGHAN Working Group on Acute Diarrhoea. Management of acute gastroenteritis in Europe and the impact of the new recommendations: a multicenter study. The Working Group on acute Diarrhoea of the European Society for Paediatric Gastroenterology, Hepatology, and Nutrition. J Pediatr Gastroenterol Nutr. 2000 May;30(5):522-7. doi: 10.1097/00005176-200005000-00011. PMID 10817282
- [Derived] Piescik-Lech M, Szymanski H, Szajewska H. Efficacy and safety of a new apple-flavoured oral rehydration solution in children with acute gastroenteritis: a double-blind randomized controlled trial. Acta Paediatr. 2012 Oct;101(10):e458-64. doi: 10.1111/j.1651-2227.2012.02782.x. Epub 2012 Aug 3. PMID 22860693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double blind, randomized controlled trial carried out in the emergency departments of 2 pediatric hospitals in Poland (The Medical University of Warsaw and St Hedvig of Silesia Hospital, Trzebnica).
Pre-assignment Details: Of the 147 children who underwent randomization, 72 were assigned to the experimental group and 75 were assigned to the control group. 17 children discontinued the study and eventually were lost to follow-up. The reason for lost to follow-up: parents refusal (N=2), not attend to scheduled visit (N=12), diarry lost (N=2), randomization error (N=1).
Groups:
- ESPGHAN ORS: ESPGHAN oral rehydration solution
  ESPGHAN ORS : Volume of the solution calculated by weight:
  * fast oral rehydration in 3-4 hours by mouth
  * ORS given for ongoing losses until diarrhea stops (maintenance phase)
- Hipp ORS Apple 200: oral rehydration solution Hipp ORS 200 Apple
  oral rehydration solution Hipp ORS Apple 200 : Volume of the solution calculated by weight:
  * fast oral rehydration in 3-4 hours by mouth
  * ORS given for ongoing losses until diarrhea stops (maintenance phase)
Period: Overall Study
Arm/Group | ESPGHAN ORS | Hipp ORS Apple 200
Started | 75 | 72
Completed | 67 | 63
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESPGHAN ORS | Hipp ORS Apple 200 | Total
Number analyzed (Participants) | 75 | 72 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 72 | 147
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.8 (0.5) | 1.6 (0.8) | 1.75 (0.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 50 | 43 | 93
Region of Enrollment [Number; unit: participants]
  Poland | 75 | 72 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Successfully Rehydrated
Description: The following components are included in primary outcome:
  * resolution of signs of dehydration
  * adequate weight gain
  * production of urine output during the trial
Time Frame: Proportion of successfully rehydrated at 24 hours
Measure: Number; unit: Participants
Arm/Group | ESPGHAN ORS | Hipp ORS Apple 200
Number analyzed (Participants) | 67 | 63
Participants | 57 | 49
Statistical Analysis 1: Comparison: Hipp ORS Apple 200; Test type: Non-Inferiority or Equivalence — The differences between study groups were considered significant when the p value was <0.05 or when the 95% CI for RD or MD did not include 0 (equivalent to p < 0.05); p = 0.28, t-test, 1 sided

2. Secondary Outcome: Unscheduled Intravenous Therapy
Description: Need for intravenous therapy within 24 hours
Time Frame: 24 hours
Measure: Number; unit: participants
Groups:
- Hipp ORS Apple 200: oral rehydration solution Hipp ORS 200 Apple
  oral rehydration solution Hipp ORS Apple 200: Volume of the solution calculated by weight:
  * fast oral rehydration in 3-4 hours by mouth
  * ORS given for ongoing losses until diarrhea stops (maintenance phase)
- ESPGHAN ORS: ESPGHAN oral rehydration solution
  ESPGHAN ORS: Volume of the solution calculated by weight:
  * fast oral rehydration in 3-4 hours by mouth
  * ORS given for ongoing losses until diarrhea stops (maintenance phase)
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
participants | 3 | 5

3. Secondary Outcome: Vomiting
Description: Vomiting starting or progressing in the first 24 hours of therapy
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
participants | 0 | 0

4. Secondary Outcome: ORS Intake in ml
Description: ORS intake in ml (in the first 24 hours, and total)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
ml | 52.4 (36.6) | 50.2 (34.6)

5. Secondary Outcome: Weight Gain in Gram
Description: Weight gain in gram (in the first 24 hours, and total)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
gram | 97 (198) | 123 (167)

6. Secondary Outcome: Duration of Diarrhea (Hrs)
Description: Time of diarrhea in hours
Time Frame: 7days
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
hrs | 69.1 (42.6) | 61.9 (38.6)

7. Secondary Outcome: Return Visit to the Emergency Department
Description: Return visit to the emergency department within a week
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
participants | 0 | 0

8. Secondary Outcome: Hospitalization
Description: need for hospitalization within a week
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
participants | 3 | 5

9. Secondary Outcome: Adverse Events
Description: any adverse event, providing a description if related or not related to study intervention
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Number analyzed (Participants) | 63 | 67
participants | 0 | 0

10. Secondary Outcome: ORS Intake at 4 h
Description: % of prescribed ORS that was consumed during first 4 hours
Time Frame: 4 hrs
Measure: Mean (Standard Deviation); unit: percentage of prescribed ORS
Arm/Group | ESPGHAN ORS | Hipp ORS Apple 200
Number analyzed (Participants) | 67 | 63
percentage of prescribed ORS | 33.6 (21) | 33.2 (24.1)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Hipp ORS Apple 200 | ESPGHAN ORS
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/67
Other Adverse Events (participants affected / at risk) | 0/63 | 0/67

LIMITATIONS AND CAVEATS:
Potential limitations included lack of perfect blinding. Because of technological reasons, it was not feasible to produce study products that were identical in colour, smell and taste.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes